CLINICAL TRIAL: NCT05094258
Title: Comparison of Early Clinical and Radiological Results and Patient Satisfaction of Mobile and Fixed Insert Unicondylar Knee Prosthesis
Brief Title: Comparison of Early Results of Mobile and Fixed Insert Unicondylar Knee Prosthesis.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Principal Investigator, Murat Sarikas, orthopaedic surgeon, Bezmialem Vakif University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 61813471876
Record Dates: First submitted 2021-10-13; First posted 2021-10-26 (Actual); Last update posted 2021-11-30 (Actual); Status verified 2021-11

CONDITIONS: Knee Osteoarthritis
Keywords: Unicompartmental Knee osteoarthritis; Unicompartmental Knee prosthesis; Mobile insert; Fixed İnsert
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Intervention Model Description: Patients with medial knee arthrosis will be randomized to receive unicompartmental knee prosthesis using mobile inserts in 30 patients and fixed inserts in 30 patients. Patients will be evaluated after at least 1 year of follow-up
Who Masked: Participant, Outcomes Assessor
Masking Description: After collecting all data about patients and patients participating in the study, the independent person who will evaluate the data will be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- mobile insert (Active Comparator): Unicondylar knee arthroplasty with mobile insert was applied to 30 patients determined by randomization. The patients were followed for 1 year.
  Interventions: Procedure: unicondylar knee prosthesis with mobile insert
- fixed insert (Active Comparator): Unicondylar knee arthroplasty with fixed insert was applied to 30 patients determined by randomization. The patients were followed for 1 year.
  Interventions: Procedure: unicondylar knee prosthesis with fixed insert

INTERVENTIONS:
Procedure: unicondylar knee prosthesis with mobile insert — Patients with unicondylar knee replacement using the mobile insert option
  Arms: mobile insert
Procedure: unicondylar knee prosthesis with fixed insert — Patients with unicondylar knee replacement using the fixed insert option
  Arms: fixed insert

SUMMARY:
Comparison of the early clinical and radiological results and patient satisfaction of the mobile and fixed insert unicondylar knee prostheses routinely used in the clinic.

DETAILED DESCRIPTION:
Unicondylar knee prosthesis operation will be performed on patients with unicompartmental knee arthrosis who apply to our clinic. Patients will be randomized to use mobile or fixed inserts. After 1 year of follow-up, SF-36, KOOS and HSS scores will be taken to examine the clinical satisfaction of the patients. In addition, radiological evaluation will be made for the presence of osteolysis at the tibial implant interface between both groups.

ELIGIBILITY:
Inclusion Criteria:

* Patients with degenerative knee arthritis with only one compartment affected

Exclusion Criteria:

* Inflammatory Arthritis
* Tricompartmental arthritis
* Patients with fixed varus deformity greater than -10 degrees
* Patients with fixed valgus deformity greater than -5 degrees
* Patients with knee range of motion less than 90 degrees
* Patients with more than 10 degrees of flexion contracture"

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-06-01 (Actual); Primary Completion 2021-12-01 (Estimated); Study Completion 2022-11-01 (Estimated)

PRIMARY OUTCOMES:
Short Form Health Survey (SF-36) | 0-1 year
  SF-36 Score (0-100) to assess patient satisfaction at postoperative 1st year
Knee injury and osteoarthritis outcome score (KOOS) | 0-1 year
  Knee injury and osteoarthritis outcome score (0-100)

CONTACTS AND LOCATIONS:
Locations (1):
- Volkan Ezici, Istanbul, Fatih, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Participant data will not be shared